CLINICAL TRIAL: NCT00759187
Title: Evaluate Clinical Research From Commerical Oral Care Products
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: William DeVizio/VP - Clinical Research, Colgate Palmolive
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CRO-0607-PLA-11-RR
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2008-11-18 (Estimated); Last update posted 2010-03-04 (Estimated); Status verified 2008-11

CONDITIONS: Gingival Diseases
MeSH Terms: conditions — Gingival Diseases | interventions — Fluorides; fluorophosphate; Triclosan; Sodium Fluoride; chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Placebo Comparator)
  Interventions: Drug: Fluoride
- B (Active Comparator)
  Interventions: Drug: Triclosan/Fluoride
- C (Active Comparator)
  Interventions: Drug: Chlorhexidine Gluconate

INTERVENTIONS:
Drug: Fluoride — Brush twice daily
  Other Names: monofluorophosphate
  Arms: A
Drug: Triclosan/Fluoride — Half mouth toothbrushing twice daily for 4 days
  Other Names: sodium fluoride; triclosan
  Arms: B
Drug: Chlorhexidine Gluconate — Mouth rinsing twice a day for 4 days
  Other Names: Chlorhexidine Gluconate oral rinse
  Arms: C

SUMMARY:
The purpose of this study is to conduct a clinical study comparing anti-plaque efficacy of commercial oral care products.

DETAILED DESCRIPTION:
The purpose of this study is to compare efficacy of two commercially available toothpastes and one oral rinse on dental plaque control.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers 18-65 years of age
* Good general health
* Must sign informed consent form
* Minimum of 20 natural uncrowned teeth (excluding third molars) must be present.
* No history of allergy to personal care consumer products, or their ingredients, relevant to any ingredient in the test products as determined by the dental/medical professional monitoring the study.

Exclusion Criteria:

* Subjects unable or unwilling to sign the informed consent form.
* Medical condition which requires pre-medication prior to dental visits/procedures
* Moderate or advanced periodontal disease or heavy dental tartar (calculus) requiring more than one visit of cleaning sessions
* 2 or more decayed untreated dental sites at screening.
* Other disease of the hard or soft oral tissues.
* Impaired salivary function (e.g. Sjogren's syndrome or head and neck irradiation).
* Use of medications that can currently affect salivary flow.
* Use of antibiotics or antimicrobial drugs within 30 days prior to study visit #1.
* Pregnant or nursing women.
* Participation in any other clinical study within 1 week prior to enrollment into this study.
* Allergy to chlorhexidine
* Use of tobacco products
* Subjects who must receive dental treatment during the study dates.
* Current use of Antibiotics for any purpose.
* Presence of an orthodontic appliance.
* History of allergy to common dentifrice ingredients.
* Immune compromised individuals (HIV, AIDS, immuno suppressive drug therapy)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Dyke, DDS, Principal Investigator
Locations (1):
- Boston University School of Dental Medicine, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Period: Overall Study
Arm/Group | Fluoride | Fluoride/Triclosan | Chlorhexidine Gluconate
Started | 8 | 8 | 9
Completed | 8 | 8 | 9
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoride | Fluoride/Triclosan | Chlorhexidine Gluconate | Total
Number analyzed (Participants) | 8 | 8 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 9 | 25
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 29.4 (6.9) | 32.6 (8.8) | 33.1 (9.0) | 31.8 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 8 | 23
  Male | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Dental Plaque Index
Description: Scale 0 to 5 (zero= no plaque to 5 = plaque covering 2/3 or more of the crown of the tooth)
Time Frame: 4-Day
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fluoride | Fluoride/Triclosan | Chlorhexidine Gluconate
Number analyzed (Participants) | 9 | 8 | 8
Units on a scale | 2.79 (0.37) | 2.82 (0.39) | 1.99 (0.41)
Statistical Analysis 1: Comparison: Fluoride vs Fluoride/Triclosan vs Chlorhexidine Gluconate; Test type: Superiority or Other; p < 0.05, ANOVA — Two way Anova general linear model (subject and treatment as factors)

ADVERSE EVENTS:
Time Frame: 4 day treatment period
Arm/Group | Fluoride | Fluoride/Triclosan | Chlorhexidine Gluconate
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/9 | 1/8 | 0/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoride (N=9) | Fluoride/Triclosan (N=8) | Chlorhexidine Gluconate (N=8)
Canker sore (General disorders) | 1 (1) | 0 (0) | 0 (0) — Aphtous lesion (canker sore) reported by patient. Patient history determined that canker sores occur after eating spicy food. Sore abated without treatment. Relationship to study product use doubtful.
Cold symptoms (General disorders) | 4 (4) | 0 (0) | 0 (0) — patient reported feeling cold symptoms. Events noted before treatment period started. Patients were on washout toothpaste (fluoride toothpaste). Relationship to study product use doubtful.
Conjunctivitis (General disorders) | 1 (1) | 0 (0) | 0 (0) — Patient reported conjuctivitis and was treated with antibiotics. Event occurred during the washout period (fluoride toothpaste) and abated after antibiotic use. Relationship to product use doubtful.
Heavy menstrual bleeding (General disorders) | 0 (0) | 1 (1) | 0 (0) — Patient reported heavy menstrual bleeding and took OTC medication and vitamins on her own. Symptoms abated after 2 days. Relationship to product use doubtful.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days